CLINICAL TRIAL: NCT05232786
Title: Awareness, Care & Treatment In Obesity Management - An Observation in Switzerland
Acronym: ACTION-CH
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-005; U1111-1266-4398 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-12; First posted 2022-02-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People / Person Living with Obesity (PLwO): From online, general population consumer panels
  Interventions: Other: No treatment given
- Health Care Professionals (HCPs): HCPs treating people who have obesity
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
ACTION Switzerland is a cross-sectional, observational, descriptive, and exploratory survey-based study without collection of laboratory data. The study is not related to any specific treatment options or pharmaceutical product. Collection of data will be performed via quantitative online survey by a third-party vendor.

The goal of this study is to provide insights to drive awareness around the needs of People Living with Obesity (PLwO) and Health Care Professionals (HCPs) involved in obesity treatment and management.

ELIGIBILITY:
Inclusion criteria:

People Living with Obesity:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male, female or other, aged above or equal to 18 years at the time of signing informed consent
3. Lives in Switzerland (minimum quota based on primary language: German, French and Italian to ensure adequate samples for sub-group analysis)
4. Current BMI of 30 Kg/m^2 or greater calculated based on self-reported height and weight

Health Care Professionals:

1. Informed consent before any study related activities (study-related activities are any procedure related to recording/collection of data according to protocol)
2. Male, female or other, aged above or equal to 18 years at the time of signing informed consent.
3. Physician
4. Dietitian who is a member of the SVDE ASDD (Swiss Association of Dietitians) and services covered by the compulsory health insurance
5. Primary Care Providers (PCPs) whose specialty is Family Practice, General Practice, General Internal Medicine (who is focused on primary care)
6. Non-PCP Specialties whose specialty is Obstetrics/Gynaecologists, Endocrinologists/Diabetologists. Psychiatrists, General Internal Medicine with focus on diabetes and/or obesity and bariatric surgeons who are involved in the management of obesity in addition to surgery
7. Practices in Switzerland
8. In clinical practice for greater than or equal to 2 years
9. Spends at least 50% time in direct patient care
10. Has seen at least 100 adult patients in past month (all physicians except psychiatrists) Has seen at least 10 patients with obesity (PCPs and General Internal Medicine with focus on Diabetes and/or obesity, Obstetrics/ Gynaecologists, Endocrinology/Diabetology or Bariatric surgery) or 5 patients with obesity (dietitians and psychiatrists) in past month needing weight management defined as: a patient with a BMI greater than or equal to 30 Kg/m^2 with or without comorbidities.

Exclusion criteria:

People Living with Obesity:

1. Previous participation in this study. Participation is defined as having given online consent in this study
2. Currently pregnant
3. Participates in intense fitness or body building programs
4. Has had significant, unintentional weight loss (due to major injury, illness, etc) in the past 6 months
5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Health Care Providers:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Unwillingness, inability, or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The respondent population will include people living with obesity (PLwO) and health care professionals (HCPs) involved in obesity treatment and management
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Weight loss motivators | At the time of survey response (Day 1)
  Multi-select from defined list
Proportion of PLwO who made serious weight loss effort | At the time of survey response (Day 1)
  Number of weight loss efforts; percentage of patients
Attitudes towards obesity and weight management and Interactions of PLwOs with HCPs | At the time of survey response (Day 1)
  5-point Likert scales (e.g., agreement, impact, frequency)
  - Proportion of responses in each category will be reported.
Weight loss barriers | At the time of survey response (Day 1)
  Multi-select from defined list
Weight loss management | At the time of survey response (Day 1)
  Multi-select from defined list

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com